CLINICAL TRIAL: NCT04955028
Title: The Application Values of MRI in Predicting Intraoperative Massive Hemorrhage for Cesarean Scar Pregnancy
Brief Title: MRI in Predicting Intraoperative Massive Hemorrhage for Cesarean Scar Pregnancy
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019442
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Cesarean Scar Pregnancy
Keywords: cesarean scar pregnancy; Ectopic pregnancy; Magnetic resonance imaging
MeSH Terms: conditions — Pregnancy, Ectopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- intraoperative massive hemorrhage: blood loss of ≥200 mL with or without artery embolization (UAE) or local CSP resection by laparoscopy or laparotomy as additional interventions.
- the non-massive hemorrhage group: blood loss of <200 mL

SUMMARY:
MRI features and clinical characteristics to predict massive hemorrhage during hysteroscopic treatment of CSP, and to aid the choice of treatment.

DETAILED DESCRIPTION:
Cesarean scar pregnancy (CSP) is a rare ectopic pregnancy occurring in cesarean section of previous cesarean delivery. The incidence of CSP was 1 in 1,800-2,216 of all deliveries reported in 2006. However, the incidence of CSP is increasing worldwide, especially in China, owing to the rapidly increasing rate of cesarean sections and second-child births since 2015.

CSP can lead to life-threatening complications, such as massive hemorrhage, uterine rupture, and loss of fertility. Therefore, immediate termination of pregnancy is recommended once a correct diagnosis is made. At present, there is still no standard treatment for CSP. Current treatments mainly include medical and surgical interventions (uterine artery embolization, suction curettage, local resection by hysteroscopy or laparoscopy, and hysterectomy). At our hospital, local resection by hysteroscopy is widely used; however, uncontrollable hemorrhage still occurs during treatment. It is of great importance to predict massive hemorrhage for clinical decision making.

Classically, transvaginal ultrasonography (TVUS) is the preferred imaging modality to diagnose CSP. However, patient factors, such as obesity, presence of bowel gas, and pain, combined with operator experience, may limit the usefulness of TVUS. Owing to excellent soft tissue contrast, the capacity of multiple dimensional images, and an excellent anatomical overview, MRI has become an important supplement to evaluate CSP and cesarean section scar (CSS). Sagittal T2-weighted imaging can be used to clearly visualize the gestational sac (GS) and the CSS of a CSP and show detailed features, including the type of CSP, the degree of CSS weakness, and the relationship between the CSP and adjacent structures. Hoffmann et al. studied 25 asymptomatic pregnant women who had undergone one previous cesarean section and found that MRI showed good inter- and intra-rater reliability in measuring lower uterine segment thickness with a low observer dependency. MRI is an additional diagnostic tool that can be used to assess the lower uterine segment in women who have undergone previous cesarean section.

To our knowledge, no previous studies have explored the relationship between MRI and intraoperative massive hemorrhage in patients with CSP. The arm of this study was to investigate the ability of clinical characteristics and MRI features to predict massive hemorrhage during hysteroscopic treatment of CSP, and to aid the choice of treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients were clinically diagnosed with CSP, which was confirmed by surgery and pathological assessment. Patients underwent local resection by hysteroscopy between January 2015 and June 2019 in our hospital. All patients underwent MRI within 3 days before surgery.

Exclusion Criteria:

* (1) twin pregnancy ; (2) preoperative methotrexate use; (3) previous incomplete CSP resection performed at other hospitals; (4) Surgical failure with incomplete CSP removal.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with Cesarean scar pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2015-01-27 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
intraoperative massive hemorrhage | intraoperative
  intraoperative blood loss

CONTACTS AND LOCATIONS:
Overall Officials: Jianyu Liu, Dr, Study Director — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No